CLINICAL TRIAL: NCT06295042
Title: The Complex Relationship of Complications and Patient-reported Outcome Measures in Autologous Versus Alloplastic Breast Reconstruction.
Brief Title: Complications and Long-term Satisfaction in Autologous vs. Implant-Based Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 32-235 ex 19/20
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Complications, Postoperative/Perioperative; Quality of Life; Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autologous Breast Reconstruction: Patients undergoing autologous breast reconstruction with free flaps
  Interventions: Other: BREAST-Q Questionnaire
- Alloplastic Breast Reconstruction: Patients undergoing alloplastic breast reconstruction with implants or expander prosthesis
  Interventions: Other: BREAST-Q Questionnaire

INTERVENTIONS:
Other: BREAST-Q Questionnaire — Patient-reported outcome measure

SUMMARY:
Current literature on complications and health-related quality of life in autologous and alloplastic breast reconstruction is inconclusive. Despite the great demand for more in-depth, long-term studies of both techniques, current evidence is low or moderate and there are only few studies focusing on both health-related quality of life and complication rates in the same patient collective.

This study aims at investigating the complex relationship between the occurrence of complications and patient-reported long-time satisfaction in autologous and alloplastic breast reconstruction.

DETAILED DESCRIPTION:
The study is conducted at the Medical University of Graz and has been approved by the responsible ethics' committee (EK: 32-235 ex 19/20). The study includes female breast cancer patients who underwent elective breast reconstruction at one of the participating departments between April 2020 and April 2023. Written informed consent was obtained from all individual study participants enrolled.

Exclusion criteria is defined as:

* Missing or insufficient information
* combination of reconstruction techniques on the same breast
* reconstruction procedures with insufficient number of cases
* inability to fully understand study procedures and to provide informed consent

Data were first collected retrospectively from the clinical data management programs using surgical reports, outpatient charts, and physicians' letters. Personal data such as patient age, concomitant diseases, nicotine abuse, anticoagulation status, previous oncological therapy and surgery, etc. were acquired. Furthermore, surgery-related data (site and type of reconstruction, size and location of implant/tissue expander, intraoperative complications) and data on the postoperative course (early and late complications, revision surgeries, number of total surgeries required, etc.) were acquired.

The five-level modified Clavien-Dindo classification is used to objectively classify postoperative complications, to allow further comparisons between treatment options, different time periods and correlations to health-related quality of life. Postoperative changes in health-related quality of life are measured using the BREAST-Q questionnaire, an effective and reliable patient-reported outcome measure in breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* female breast cancer patient undergoing autologous or alloplastic breast reconstruction willing to participate in this study
* age between 18 and 80 years (upper limit due to indication for breast reconstruction)
* written informed consent

Exclusion Criteria:

* Missing or insufficient information
* combination of reconstruction techniques on the same breast
* reconstruction procedures with insufficient number of cases
* inability to fully understand study procedures and to provide informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients between 18 and 80 years who underwent autologous or alloplastic breast reconstruction at our department, willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Complications | Retrospective data analysis at the time of study inclusion (up to 10 years postoperative)
  The five-level modified Clavien-Dindo classification is used to objectively classify postoperative complications. A subgroup analysis will be done for complications requiring revision surgery under general anesthesia and complications not requiring revision surgery under general anesthesia.

SECONDARY OUTCOMES:
Health-related quality of life and satisfaction | Retrospective data analysis at the time of study inclusion (up to 10 years postoperative)
  Postoperative changes in health-related quality of life are measured using the BREAST-Q questionnaire (postoperative, reconstructive module), an effective and reliable patient-reported outcome measure in breast reconstruction. Questions in each category can be answered on a scale from 0 to 100, with 100 indicating the highest satisfaction or well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis